CLINICAL TRIAL: NCT04702100
Title: Instrument-assisted Soft Tissue Mobilization Versus Integrated Neuromuscular Inhibition Technique on Mechanical Non-specific Neck Pain
Brief Title: Instrument-assisted Soft Tissue Mobilization Versus Integrated on Mechanical Neck Pain
Acronym: IASTM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Al Shaymaa Shaaban Abd El Azeim, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: p.t.REC/012/003038
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Non-specific Chronic Mechanical Neck Pain
Keywords: instrument-assisted soft tissue mobilization; integrated neuromuscular inhibition technique

STUDY DESIGN:
Intervention Model Description: instrument assisted soft tissue mobilization and integrated neuromuscular inhibition technique
Who Masked: Participant, Outcomes Assessor
Masking Description: random generator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- instrument assisted soft tissue mobilization (Experimental): the patients will receive instrument-assisted soft tissue mobilization+conventional therapy three times per week for four week
  Interventions: Other: instrument assisted soft tissue mobilization; Other: conventional therapy
- integrated neuromuscular inhibition technique (Experimental): the patients will receive integrated neuromuscular inhibition technique+ conventional therapy. three times a week for four week
  Interventions: Other: integrated neuromuscular inhibition technique; Other: conventional therapy
- conventional therapy (Active Comparator): the patients will receive conventional therapy three times a week for four week
  Interventions: Other: conventional therapy

INTERVENTIONS:
Other: instrument assisted soft tissue mobilization — the patients will receive instrument-assisted soft tissue mobilization:The subject was seated in a relaxed sitting position. M2T blade was used to find specific areas of restriction on RT upper trapezius. Then treatment plane 1 - 2 and 3 were used.The lubricant (Vaseline) was applied to the skin around the neck area prior to treatment and the tool was cleaned with an alcohol preparation pad. Then by using M2T blade with angle 45, we were giving long slow strokes without causing any discomfort or pain over muscle starting from its insertion up to its origin approximately for 2 to 3 min repeated two times.
  Arms: instrument assisted soft tissue mobilization
Other: integrated neuromuscular inhibition technique — will receive integrated neuromuscular inhibition technique: from supine lying position.we the patients will perform ischemic compression at trigger points then positional release technique and finally muscle energy technique.
  Arms: integrated neuromuscular inhibition technique
Other: conventional therapy — the patients will receive hot back for 10 minutes, active range of motion exercise, chin tuck, stretches

SUMMARY:
the aim of this study is to investigate the efficacy of instrumented assisted soft tissue mobilization versus integrated neuromuscular inhibition technique on mechanical non-specific neck pain

DETAILED DESCRIPTION:
Mechanical neck pain is a prevalent condition in various populations. Neck pain occurrence is affected by several factors, involving environmental, psychological, and social aspects. Neck pain represents the fourth major disorder responsible for a person's year lived with disability and ranked eleventh as disability-adjusted life years of a person. The neck pain incidence ranges from 10.4 to 23.3% in 1-year time, while the range of prevalence was 0.4 to 86.8%. It has a high prevalence among computer users, office workers, and females, especially females aged 35 to 49 years old. Myofascial trigger point (MTrP) might play an important role in the formation of mechanical neck pain and is known as a hyperirritable spot in skeletal muscle that is accompanied with a hypersensitive palpable nodule in a taut band. IASTM and integrated play an important role in the treatment of mechanical neck pain.this trial has three groups; one will receive IASTM+ conventional, the second will receive integrated + conventional and the third will receive conventional treatment for four week

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed as non-specific neck pain with upper trapezius active myofascial trigger points less than 3 months of duration and have these criteria: taut band on palpation, hyper sensible tender spot in the taut band, local twitch response referred pain pattern
2. body mass index from 18 to 25 kg/m2
3. their ages from 18-35

Exclusion Criteria:

1. if they had trigger point injections within the past 6 months
2. history of neck or upper back surgery, trauma or fracture
3. history of a whiplash injury, skin diseases and lesions, any sensory disturbances, any vascular syndromes, neck and back deformities
4. cervical radiculopathy, and diagnosis of fibromyalgia syndrome, skin diseases

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
pain intensity | up to four weeks
  The scale that will be used the VAS ;each subject will instructed to put point on line from no pain to tolerable pain

SECONDARY OUTCOMES:
neck disability | up to four weeks
  will be measured by Arabic neck disability index
muscle amplitude in the form of normalized root mean square (RMS) | up to four weeks
  muscle amplitude will be measured by surface electromyography for upper trapezius
muscle fatigue in the form of median frequency | up to four weeks
  muscle fatigue will be measured by surface electromyography for upper trapezius

CONTACTS AND LOCATIONS:
Locations (1):
- Al Shaymaa Shaaban Abd El Azeim, Giza, Egypt